CLINICAL TRIAL: NCT02554669
Title: Acute Effects of Postabsorptive and Postprandial Physical Activity on Glycemia and Inflammation
Brief Title: Acute Effects of Postabsorptive and Postprandial Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: papa vs pppa
Record Dates: First submitted 2015-05-23; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Hyperglycemia; Inflammation
Keywords: Blood glucose (indicated by interstitial glucose); Markers of systemic inflammation
MeSH Terms: conditions — Hyperglycemia; Inflammation | interventions — Postprandial Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No physical activity
- Postabsorptive physical activity (Experimental): Physical activity performed before breakfast
  Interventions: Behavioral: postprandial and postabsorptive physical activity on treadmill
- Postprandial physical activity (Experimental): Physical activity performed in the postprandial period after breakfast
  Interventions: Behavioral: postprandial and postabsorptive physical activity on treadmill

INTERVENTIONS:
Behavioral: postprandial and postabsorptive physical activity on treadmill
  Arms: Postabsorptive physical activity; Postprandial physical activity

SUMMARY:
Physical activity performed in the postprandial state has the ability to blunt postprandial glycemia acutely, even as a result of very light or small amounts of postprandial physical activity. Postprandial physical activity decreases postprandial glycemia more effectively than activity performed in the post-absorptive state. However, studies comparing postprandial and postabsorptive physical activity have measured glycemic outcomes in only short periods of time (hours) or have used a very large dose of physical activity.

Physical activity have the ability to entail an acute increase in markers of systemic inflammation.Previous studies has also shown that systemic inflammation is increased during glycemic spikes, such as after a high carbohydrate load. Therefore the effect of postprandial physical activity is difficult to predict. One one hand it might increase markers of systemic inflammation. On the other hand it might decrease systemic inflammation as a result of a blunting effect on postprandial glycemia. The effect of physical activity after carbohydrate intake might therefore also differ from postabsorptive physical activity.

Purpose of the study: I) The investigators hypothesized that light physical activity performed in the post-prandial sate decrease blood glucose in a day and night cycle compared to the same activity performed in the postabsorptive state and a control day. II) To test whether postabsorptive and postprandial light physical activity do affect markers of systemic inflammation different.

12 participants diagnosed with hyperglycemia but not on hypoglycemic medication took part in a randomized cross-over trial with 3 test days. A control day with no physical activity, and two days similar to the control day except that one of them contained a one hour bout of treadmill walking prior to breakfast and the other a similar exercise bout after breakfast. Continuous glucose monitoring was performed from start of exercise / breakfast until the morning next day (at least 22 hours). Venous blood was also sampled at given timepoints (before exercise / before breakfast, and 1.5, 2.5, 3.5 and 24 hours after breakfast. Dietary intake was individually standardized prior to and during test days.

DETAILED DESCRIPTION:
Physical activity performed in the postprandial state has the ability to blunt postprandial glycemia acutely, even as a result of very light or small amounts of postprandial physical activity. Postprandial physical activity decreases postprandial glycemia more effectively than activity performed in the post-absorptive state. However, studies comparing postprandial and postabsorptive physical activity have measured glycemic outcomes in only short periods of time (hours) or have used a very large dose of physical activity.

Physical activity have the ability to entail an acute increase in markers of systemic inflammation.Previous studies has also shown that systemic inflammation is increased during glycemic spikes, such as after a high carbohydrate load. Therefore the effect of postprandial physical activity is difficult to predict. One one hand it might increase markers of systemic inflammation. On the other hand it might decrease systemic inflammation as a result of a blunting effect on postprandial glycemia. The effect of physical activity after carbohydrate intake might therefore also differ from postabsorptive physical activity.

Purpose of the study: I) The investigators hypothesized that light physical activity performed in the post-prandial sate decrease blood glucose in a day and night cycle compared to the same activity performed in the postabsorptive state and a control day. II) To test whether postabsorptive and postprandial light physical activity do affect markers of systemic inflammation different.

12 participants diagnosed with hyperglycemia but not on hypoglycemic medication took part in a randomized cross-over trial with 3 test days. A control day with no physical activity, and two days similar to the control day except that one of them contained a one hour bout of treadmill walking prior to breakfast and the other a similar exercise bout after breakfast. Continuous glucose monitoring was performed from start of exercise / breakfast until the morning next day (at least 22 hours). Venous blood was also sampled at given timepoints (before exercise / before breakfast, and 1.5, 2.5, 3.5 and 24 hours after breakfast. Dietary intake was individually standardized prior to and during test days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hyperglycemia

Exclusion Criteria:

* Use of hypoglycemic agents or diseases directly affecting blood glucose, except of diabetes type 2 / insulin resistance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in interstitial glucose from test day to test day | Measured continuously on each test day, but a mean of every 5. minute during test day (from breakfast until 22 hours after breakfast) is stored and used for analysis (acute effect in a cross-over design).
  Interstitial glucose, measured by continuous glucose monitoring
Change in hsCRP from test day to test day | Measured on each test day (acute effect in a cross-over design). A mean of the samples before exercise / before breakfast, and 1.5, 2.5, 3.5 and 24 hours after breakfast is used for analysis of change from test day to test day
  This is a marker of inflammation, it will be measured from plasma of venous blood samples
Change in VCAM from test day to test day | Measured on each test day (acute effect in a cross-over design). A mean of the samples before exercise / before breakfast, and 1.5, 2.5, 3.5 and 24 hours after breakfast is used for analysis of change from test day to test day
  This is a marker of inflammation, it will be measured from plasma of venous blood samples

SECONDARY OUTCOMES:
Change in Blood glucose (venous samples) from test day to test day | Measured on each test day (acute effect in a cross-over design). A mean of the samples before exercise / before breakfast, and 1.5, 2.5, 3.5 and 24 hours after breakfast is used for analysis of change from test day to test day
  Plasma samples of venous blood
Change in triglycerides from test day to test day | Measured on each test day (acute effect in a cross-over design). A mean of the samples before exercise / before breakfast, and 1.5, 2.5, 3.5 and 24 hours after breakfast is used for analysis of change from test day to test day
  Plasma samples of venous blood

OTHER OUTCOMES:
Change in oxygen consumption from test day to test day | Measured on each test day (acute effect in a cross-over design). A mean of the samples during exercise, and 1, 2 and 3 hours after breakfast is used for analysis of change from test day to test day
  Measured by indirect calorimetry
Change in heart rate from test day to test day | Measured on each test day (acute effect in a cross-over design). A mean of the samples during exercise, and 1, 2 and 3 hours after breakfast is used for analysis of change from test day to test day
  Measured by a heart rate sensor
Change in lactic acid from test day to test day | Measured on each test day (acute effect in a cross-over design). A sample after 59 minutes of exercise is used for analysis of difference between intervention days
  measured from capillary finger sticks
Change in Respiratory exchange ration (RER) from test day to test day | Measured on each test day (acute effect in a cross-over design). A mean of the samples during exercise, and 1, 2 and 3 hours after breakfast is used for analysis of change from test day to test day
  Measured by indirect calorimetry